CLINICAL TRIAL: NCT05448352
Title: The APPLE Study; a Cross-sectional Study Exploring Diet, Life-style Patterns and Psoriasis Severity
Brief Title: Asking People With Psoriasis About Lifestyle and Eating
Acronym: APPLE
Status: Completed | Type: Observational
Sponsor: King's College London (Other)
Collaborators: Psoriasis Association (Unknown)
Responsible Party: Sponsor
Other Study IDs: Worktribe ref 1121143
Record Dates: First submitted 2022-06-14; First posted 2022-07-07 (Actual); Last update posted 2024-01-26 (Actual); Status verified 2023-06

CONDITIONS: Psoriasis
Keywords: Diet; Lifestyle; Sleep; Physical Acitivty; Wellbeing
MeSH Terms: conditions — Psoriasis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The APPLE Study aims to understand if specific diet and lifestyle patterns are present in individuals with psoriasis and if these factors are correlated with psoriasis severity.

DETAILED DESCRIPTION:
Prospective participants will be invited to read an information sheet and provide informed consent. Once informed consent is obtained, participants will be screened for eligibility with a short online screening questionnaire. Upon successful completion, participants will be directed to start the online multiple-choice survey with questions on psoriasis, diet and lifestyle patterns and complete a 4-day diet diary.

ELIGIBILITY:
Inclusion Criteria:

Adults (18 years of age or older) Dermatologist diagnosis of psoriasis Residents in the United Kingdom (UK) Fluent in English

Exclusion Criteria:

Minors (17 years of age or younger) Not medically diagnosed with Psoriasis Non-UK residents

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population will comprise of adults, with a medical diagnosis of psoriasis living in the UK and who are fluent in the English language. This is a nationwide study to obtain responses from participants representative of the psoriasis population in the UK.
Sampling Method: Non-Probability Sample
Enrollment: 358 (Actual)
Dates: Start 2022-06-18 (Actual); Primary Completion 2024-01-08 (Actual); Study Completion 2024-01-08 (Actual)

PRIMARY OUTCOMES:
self-assessed Simplified Psoriasis Index | Baseline
  The self-assessed Simplified Psoriasis Index measures psoriasis severity as a joint score of 3 categories.
  Severity; a 3-point scale will measure the severity of skins lesions on 10 body parts. 0=minimal, +/-=noticeable. + =extensive. A 5-point scale ranging from 0=clear to 5=intensely inflamed skin will measure the overall state of psoriasis.
  Psychosocial; a 10 point scale ranging from 0=not at all to 10=very much will indicate the extent to which psoriasis is affecting day-to-day life.
  Intervention; participants will need to indicate each psoriasis treatment that is being received. 1 point per treatment.
  The sa-PSI will generate a total score out of 70. The higher the score, the greater the severity of psoriasis.
The Dermatology Life Quality Index (DLQI) | Baseline
  This index measures the impact of psoriasis on day-to-day routines as well as on psychological and social fronts. Responses to questions are scored as follows: very much (3 points), a lot (2 points), a little (1 point), not at all/not relevant (0 points).
  The DLQI provides a score between 0-30. The score range is interpreted as follows: 0-1 points = no effect at all on the participants life, 2-5 points = small effect on participant's life, 6-10 points = moderate effect on participant's life, 11-20 = very large effect on participant's life and 21-30 = extremely large effect on participant's life.
Diet | Baseline
  The Twins United Kingdom (TwinsUK) modified European Prospective Investigation into Cancer Food Frequency Questionnaire (EPIC FFQ) will assess dietary intake.
  This FFQ will provide an overview of the consumption of 131- food items over the past 12 months. Each food item will be rated on a 9 point scale as follows: Never or less than once a month, 1-3 times per month, Once a week, 2-4 per week, 5-6 per week, Once a day, 2-3 per day, 4-5 per day and 6+ per day.
Diet | 4 day 24-hour dietary recall
  Nutrient consumption will be examined using the Intake24 (https://intake24.co.uk/). This is dietary assessment tool in which participants will record their food intake over the past 24 hours. The results obtained from the Intake24 will provide a detailed breakdown of the total calories, macronutrients and micronutrients consumed.

SECONDARY OUTCOMES:
Sleep | Baseline
  Questions from the Pittsburgh Sleep Quality Index will be used to evaluate sleep quality, latency and duration.
  Sleep quality: is measured on a 4-point scale ranging from very bad to very good.
  Sleep latency: participants will indicate the number of minutes taken to fall asleep on a weekday and weekend day. The 6-point scale ranges from 0-10 minutes to 60+ minutes.
  Sleep duration: participants will indicate the number of hours of actual sleep that are obtained on a weekday/weekend day.
Physical Activity (PA) | Baseline
  The International Physical Activity Questionnaire (IPAQ) categorises PA into vigorous intensity, moderate intensity and walking. The frequency (number of days/week) and the duration (number of hours) for each PA category will determine the participant's PA level:
  Health Enhancing Physical Activity (HEPA)=vigorous intensity physical activity is undertaken on at least 3 days/ week with a minimum of 1500 metabolic equivalent (MET) minutes/week or with 7 or more days of any combination of walking, moderate or vigorous intensity activities with a minimum of 3000 MET minutes/week.
  Minimally active (any one of the following)=3 or more days of vigorous activity with at least 20 minutes/day, 5 or more day of moderate intensity or walking at least 30 minutes/day, or 5 or more days of combination of walking, moderate or vigorous intensity activities with a minimum of 600 MET minutes/week.
  Inactive=no activity is reported or if some activity is reported but does not meet the above criteria.
Alcohol | Baseline
  The frequency and units of alcohol intake will be examined using the Alcohol Use Disorders Identification Test Consumption (AUDIT-C).
Smoking | Baseline
  Smoking status will be evaluated as smoker, non-smoker or ex-smoker.
Meal timings | Baseline
  Meal timings will be captured using the Food Timing Questionnaire.
Demographic characteristics | Baseline
  The demographic characteristics assessed include age, gender and ethnicity.
General Health | Baseline
  General health will be examined based on the presence of health conditions such as obesity, cardiovascular disease, diabetes etc.
Dietary habits | Baseline
  Dietary habits will be evaluated based on the inclusion and exclusion of food items from diet, beliefs around diets and following specific diets as means to improve psoriasis.

CONTACTS AND LOCATIONS:
Locations (1):
- King's College London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2022-05-30): https://cdn.clinicaltrials.gov/large-docs/52/NCT05448352/ICF_000.pdf